CLINICAL TRIAL: NCT04929925
Title: The Role of Serum Procalcitonin in Diagnosis and Detection of Outcome of Acute Bacterial Meningitis in Children.
Brief Title: The Role of Serum Procalcitonin in Diagnosis and Detection of Outcome of Acute Bacterial Meningitis in Childern
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Marina Wahib Shawky, resident doctor at pediateric department sohag university hospital, Sohag University
Other Study IDs: Soh-Med-21-04-01
Record Dates: First submitted 2021-04-14; First posted 2021-06-18 (Actual); Last update posted 2021-06-18 (Actual); Status verified 2021-04

CONDITIONS: CNS Infection in Children
Keywords: Serum procalcitonim

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: serum procalcitonin in acute bacterial meningitis — Serum Procalcitonin estimation will be done by Cobas e411Roch diagnostic,Switzerland apparatus by immunoassay method (electrochemiluminescence immunoassay) by using sample serum or plasma heparin or EDTA with reference range less than 0.5ng/ml ( no sepsis) but 0.5-2ng/ml)follow up is recommended) and more than 2 (sepsis)

SUMMARY:
Meningitis is one of the most common central nervous system (CNS) infections encountered in infants and children. The source of infection in meningitis can be bacterial, viral, fungal, or parasitic in origin . Bacterial meningitis is a paediatric emergency with high mortality and morbidity rate. Hence it must be diagnosed and treated promptly. But the similar clinical presentation often makes it difficult to differentiate bacterial and non-bacterial aetiologies in children .

DETAILED DESCRIPTION:
Meningitis is one of the most common central nervous system (CNS) infections encountered in infants and children. The source of infection in meningitis can be bacterial, viral, fungal, or parasitic in origin . Bacterial meningitis is a paediatric emergency with high mortality and morbidity rate. Hence it must be diagnosed and treated promptly. But the similar clinical presentation often makes it difficult to differentiate bacterial and non-bacterial aetiologies in children .

Currently, cerebrospinal fluid (CSF) analysis has been considered the gold standard for diagnosing bacterial meningitis, along with biomarkers like C-reactive protein (CRP) and white blood cell count (WBC) . However, clinical criteria, gram staining, and bacterial antigen testing of CSF as well as the classic biological markers in blood (CRP, WBC, and neutrophil count) or CSF (protein level, glucose level, WBC, and neutrophil count) used alone do not offer 100% sensitivity and specificity for distinguishing bacterial and non-bacterial meningitis .Moreover, two or more days of waiting is required to identify bacterial growth in CSF cultures Procalcitonin, a 116-amino-acid peptide, which undergoes posttranslational proteolysis into calcitonin, is synthesized in C cells of the thyroid gland and secreted from leukocytes of the peripheral blood. The level of PCT increases (without an increase in calcitonin level) in the presence of bacterial lipopolysaccharides and cytokines that are associated with severe bacterial infections . In contrast to this, there is minimal rise of PCT in patients infected with viruses . Moreover, there is dramatic and quick increase in serum PCT levels after a single endotoxin injection . This type of response to a bacterial stimulus makes PCT level a potentially sensitive marker of severe bacterial infections including meningitis.

After intensive research for new and rapid diagnostic methods for differential diagnosis of meningitis, serum procalcitonin (PCT) has been demonstrated to be the best marker for diagnosis of sepsis that also correlates with the extent and severity of microbial invasion . Procalcitonin is now considered to be clinically most useful and superior to CRP due to its high diagnostic accuracy in various infectious pathologies, including sepsis, acute infectious endocarditis, and pancreatitis .Several studies have demonstrated the raised values of serum PCT in bacterial infections including meningitis . Studies from adults have shown PCT as a powerful diagnostic test for the assessment of suspected meningitis, allowing rapid differentiation between bacterial and non-bacterial (mostly viral) aetiologies, and earlier initiation of appropriate and necessary therapies. The evidence suggests that while serum PCT offers a similar specificity to the traditionally used CSF markers of meningitis, it also confers a higher sensitivity allowing for a more accurate overall diagnosis in patients with suspected meningitis.

There is a little studies on the role of serum procalcitonin in the diagnosis and prognosis of acute bacterial meningitis in children

ELIGIBILITY:
Inclusion Criteria:

* All children from one month of age to 14 years old with confirmed and full filling the diagnostic criteria of meningitis .
* Cases: children surely diagnosed with acute bacterial meningitis .
* Controls: children with suspected non-bacterial meningitis .

Exclusion Criteria:

* neonates
* children with other systemic or focal infections
* children with other neurological problems(CNS hemorrhage or infarction, epilepsy and other causes of convulsions, cerebral palsy and other neurodegenerative and metabolic diseases)

Ages: 1 Month to 14 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Study Population: Children with CNS infection from one month to 14 years
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2021-06-15 (Estimated); Primary Completion 2022-07-15 (Estimated); Study Completion 2022-07-15 (Estimated)

PRIMARY OUTCOMES:
To asses the serum level of procalcitonin diagnosis of acute baterial meningitis in children | one year
  * to study the role of serum procalcitonin in diagnosis and differentiation of acute bacterial from non-bacterial causes of meningitis.
  * with refrance range :
  * Less than .5ng/ml (no sepsis )
  * (.5 -2ng/ml ) (follow up is recommended) .
  * more than 2 ng /ml (sepsis )

IPD SHARING:
Plan to Share IPD: Undecided
undecided